CLINICAL TRIAL: NCT03729973
Title: Comparing The Efficacy Of Preoperative Nebulized: Ketamine, Magnesium Sulfate, and Lidocaine In Attenuating Postoperative Sore Throat After Endotracheal Intubation
Brief Title: Comparing Efficacy Preoperative Nebulized: Ketamine , Mgspo4 ,and Lidocaine In Attenuating Endotracheal Sore Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Alshaimaa Abdel Fattah Kamel, lectuerer, Zagazig University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 4915
Record Dates: First submitted 2018-10-27; First posted 2018-11-05 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Sore Throat
MeSH Terms: conditions — Pharyngitis | interventions — Ketamine; Magnesium Sulfate; Lidocaine; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (K) (Active Comparator): Group (K) (n=25): patients nebulized ketamine 50 mg(milgram) (1ml) plus 4ml normal saline.So total volume (5ml).
  In preparation room an I.V line was secured ,and stranded monitoring was connected to patient.
  Patients nebulized 1ml ketamine (Ketalar 50mg/VI Solution for Injection) by compressor nebulizing for 15 minutes.
  Interventions: Drug: Ketamine
- Group (M) (Active Comparator): Group M(n=25) : patients nebulized isotonic magnesium sulfate 250mg (3ml)( 50% Magnesium Sulfate Injection)plus 1ml normal saline.
  In preparation room an I.V line was secured ,and stranded monitoring was connected to patient.
  Patients nebulized by compressor nebulizing for 15 minutes.
  Interventions: Drug: Magnesium Sulfate
- Group (L) (Active Comparator): Group (L) (n=25): patients nebulized lidocaine 2% 100mg .So total volume (5ml). In preparation room an I.V line was secured ,and stranded monitoring was connected to patient.
  Patients nebulized by compressor nebulizing for 15 minutes.
  Interventions: Drug: Lidocaine
- Group (C) (Active Comparator): Group (C) (n=25): patients nebulized normal saline(0.9%). 5ml .In preparation room an I.V line was secured ,and stranded monitoring was connected to patient.
  Patients nebulized by compressor nebulizing for 15 minutes.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine — Patients nebulized ketamine by compressor nebulizing for 15 minutes.
  Other Names: (Ketalar, 50 Mg/mL Injectable Solution)
  Arms: Group (K)
Drug: Magnesium Sulfate — Patients nebulized magnesium sulfate 250mg (3ml)plus 2ml normal saline by compressor nebulizing for 15 minutes.
  Other Names: (Magnesium Sulfate 500 /ML)
  Arms: Group (M)
Drug: Lidocaine — In preparation room an I.V line was secured ,and standard monitoring was connected to patient.
  Patients nebulized lidocaine 5ml by compressor nebulizing for 15 minutes.
  Other Names: (Xylocaine 2 % Injectable Solution)
  Arms: Group (L)
Drug: Normal saline — In preparation room an I.V line was secured ,and standard monitoring was connected to patient.
  Patients nebulized by compressor nebulizing 5ml normal saline for 15 minutes.
  Other Names: (Normal Saline 0.9% Infusion Solution)
  Arms: Group (C)

SUMMARY:
One of the most common complications after endotracheal intubation is sore throat Lidocaine jelly or spray, preoperative gargles with licorice or ketamine or I.V steroids used for prophylaxis against POST are expensive ,and having much more side effects,but nebulized lidocaine is easily found with decreasing cost ,easily administered ,acts immediately with short duration ,minimal side effects ,and no term residual side effects.

Nebulized ketamine was found to have a protective effect on allergen-induced airway inflammatory injury , high airway reactivity ,and decreasing postoperative sore throat (POST) incidence .

Magnesium sulfate is similar to ketamine in blocking the N-methyl-D-aspartate receptors.

DETAILED DESCRIPTION:
Patients and Methods a) Sample size:Assuming that mean+standard Deviation of age of nebulized ketamine group is 42.3+11.9 and normal saline group is 35.5+11.7 .So sample size is calculated by open source Epidemiologic statistics for public health (openEpi) to be 100 cases in 4 groups (25 cases in each group) with confidence level 95% and power of test is 80%.

All Cases Will Undergo:

a. Patient Examination: All participating patients will be interviewed preoperatively during their preoperative preparation. The goal and endpoints of the study will be discussed. and written informed consent will be included in the study.

On physical examination, special attention will be given to document vital signs, cardiac, chest condition and exclude exclusion criteria , laboratory investigations will be reviewed ..

In preparation room an I.V line was secured ,and stranded monitoring was connected to patient.

Patients nebulized by compressor nebulizing for 15 minutes. Patient was then transferred to operating room where a stranded monitor was connected (Non-invasive blood pressure, pulse oximeter, ECG,and capnography).

Patient was pre-oxygenated with 5 Litter/min (L/min) O2, 100% for 3-5 min. premedication with glycopyrrolate 0.01 milgram/kilogram (mg/kg), midazolam 0.02mg/kg.

Induction was done by fentanyl 2ug/kg, propofol 2mg/kg, endotracheal intubation was facilitated by atracurium 0.6mg/kg, and intubation by soft seal cuffed sterile polyvinyl chlorid tracheal tube of 7mm inner diameter in female ,and 8mm in male patients, the cuff was inflated with air.All intubation was performed by an experienced anaesthesiologist.

Maintenance of anaesthesia done using isoflurane 1 Minimum Alveolar Concentration (MAC) ,and atracurium. The last dose of atracurium was given 20 min. before extubation.

At the end of the surgery, the inhalational anaesthetic was turned off, and the muscle relaxant was reversed by a combination of neostigmine 0.05mg/kg, and glycopyrrolate 0.01mg/kg.The patient was extubated after extubation criteria were met, and the patient was transferred to recovery room.

In the recovery room, all patients received O2 2.5L/min by face mask.The presence of sore throat was noted at rest and on swallowing immediately after extubation.

The intensity of sore throat was recorded at 2,4,8,12,24 hours postoperatively. In postoperative ward, patients were also monitored haemodynamics (BLp, O2 saturation, pulse), drug related side effects,and sedation level using A=Alert, V=Verbal, P=Painful,U=Unresponsive ( AVPU)score .

Sore throat was measured on 4 point scale (0-3). 0= no sore throat

1. mild sore throat (complaint of sore throat on asking).
2. moderate sore throat (change in voice or hoarseness associated with throat pain).
3. sever sore throat (change in voice or hoarseness associated with throat pain). Protocol for pain management, I.V diclofenac 75mg every 12h. Patient with sore throat score = 2 or 3 will be treated with IV diclofenac 1mg/kg every 8h.

Patient satisfaction:The patients will be asked to rate the overall degree of satisfaction of the analgesia using a 1-3 verbal scale (1 = unsatisfactory analgesia, 2 = satisfactory analgesia, and 3 = excellent analgesia) .

VII- Side effects and Complications as: Nausea, Vomiting, Local anaesthetics toxicity or other complications will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age (21-45) years old.
* American Society of Anesthesiologists (ASA) I / II
* elective surgery of approximately 2-3h duration needing endotracheal intubation
* Patient With BMI(Body Mass Index)(25-30)

Exclusion Criteria:

* Patient refusal.
* Altered mental status.
* History of allergy to drugs in the study
* .Patients with history of pervious sore throat
* using steroids or NSAIDs,with asthma
* neuromuscular disease
* , Mallampati grade>2, with >2 attempts of intubations,
* underlying neck ,and laparoscopic surgeries,
* pregnant women.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
4 point sore throat intensity: self reported sore throat intensity at 2,4,8,12,24 hours postoperatively. . | 2,4,8,12,24 hours
  The intensity of sore throat will be recorded at 2,4,8,12,24 hours postoperatively on 4 point scale (0-3):
  0= no sore throat
  1. mild sore throat (complaint of sore throat on asking).
  2. moderate sore throat (change in voice or hoarseness associated with throat pain).
  3. sever sore throat (change in voice or hoarseness associated with throat pain).

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Kamel, MD, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University Hospitsals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No